CLINICAL TRIAL: NCT02081638
Title: Elite Controller and ART-Treated HIV+ Statin Versus ASA Treatment Intervention Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140039; 14-I-0039
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: Treated Progressors; Immune Activation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Aspirin; Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elite Controller (Active Comparator): Elite controllers not on ART
  Interventions: Drug: Aspirin; Drug: Atorvastatin
- Treated Progressors (Active Comparator): HIV infected on ART
  Interventions: Drug: Aspirin; Drug: Atorvastatin

INTERVENTIONS:
Drug: Aspirin — Daily Asprin daily
Drug: Atorvastatin — Daily Atorvastatin Daily

SUMMARY:
Background:

- The immune system protects the body from infection. But it can also cause harm. For example, the clotting system makes blood clot and protects from bleeding. But blood clots are sometimes harmful. People with human immunodeficiency virus (HIV) infection have increased inflammation and clotting. This may increase their risk for diseases like stroke or heart attack. Researchers want to know how aspirin or HMG-CoA reductase inhibitors (so-called statin medications) affect the immune and clotting systems of people with HIV. Aspirin is a medicine to decrease clotting. Statins are medications given to lower cholesterol and decrease inflammation.

Objectives:

- To see how aspirin or statins change immune and clotting systems in people with HIV.

Eligibility:

- Adults 18 and older with HIV and a low viral load, not on aspirin or a statin medication. They must also have either: (1) never taken anti-HIV medications (ARVs), have a suppressed viral load, have stable CD4 counts, and never had an opportunistic infection; or (2) been taking ARVs for 5 continuous years and have a suppressed viral load for more than 3 years.

Design:

* Participants will be screened with medical history, physical exam, and blood and lab tests.
* Participants will repeat screening tests and have an MRI. An MRI is a way to visualize blood vessels in the neck and head. Participants will lie on a table that slides in and out of a cylinder surrounded by a magnetic field.
* Participants will take either study drug once daily for 9 months.
* Participants will have a blood procedure twice. Blood will be removed through a needle in one arm and circulated through a machine that removes white blood cells. The blood, minus white blood cells, is returned through a needle in the other arm.
* All participants will be observed for 3 months before and after treatment.

DETAILED DESCRIPTION:
Despite dramatic improvements in mortality with antiretroviral therapy (ART), HIV-infected persons remain at risk of developing non-infectious complications, including cardiovascular, renal, and neurological disease. A small subset of the HIV-infected population achieve durable control of HIV virus in the absence of ART. These individuals, termed elite controllers (ECs), remain ART na(SqrRoot) ve, have stable CD4 T cell counts for many years and have no history of opportunistic infections. Despite the lack of AIDS complications, recent evidence suggests ECs may exhibit heightened immune activation that may contribute to a potentially increased risk for non-infectious complications, similar to successfully treated progressors.

In the current 2 group, randomized, open label trial, we intend to study the effects of a lipid lowering agent vs aspirin (ASA) on immune activation in HIV-1 infected participants. One group will consist of ECs who are HIV-1 infected, maintain HIV-RNA levels of less than the LLD of commercially available assays in the absence of ART, have no history of ART or opportunistic infections (OIs) and have stable CD4 T cell counts for greater than 3 years. The second group will enroll HIV-1 infected Treated Progressors (henceforth referred to as ART <50) who have maintained HIV-RNA below the limit of detection in commercially available assays (<40, <48, or <50 copies/mL) for greater than 3 years on ART (treatment duration greater than 4 years). Up to 2 months after the screening and enrollment visit, each group will enter a 3 month observation period (to establish baseline values for biomarkers/cellular markers). After 3 months, participants from each group will be randomized to either ASA, 81 mg PO daily, or atorvastatin (ATV), 40 mg (dose adjusted for subjects on antiretroviral regimens with significant interactions, and will be treated for 9 months, followed by 3 months of a wash out period (see Figure 1). The primary end point will be change of sCD14 after 9 months of study intervention from Month 3 to Month 12 in each treatment arm, with groups combined (EC and ART <50). Secondary objectives will be to compare changes in soluble biomarkers (sCD14, IL-6, D-dimer, hsCRP, sTF, sCD163 and other relevad treatment arms (ASA vs statin and EC vs ART<50 and with groups combined), to evaluate cardiovascular (CV) disease prevalence in EC vs ART<50 and with groups combined), to evaluate cardiovascular (CV) disease prevalence in EC vs ART <50 by MR imaging of carotids, to determine MR measurements and correlations with biomarkers and cellular activation markers, and to investigate changes in plasma viremia as measured by single copy assay over time.

ELIGIBILITY:
* INCLUSION CRITERIA:

EC Arm

1. Age greater than or equal to 18 years.
2. Documented HIV-1 infection confirmed by enzyme-linked immunosorbent assay (ELISA) and Western blot tests (will not be repeated if performed previously at NIH).
3. Categorized as a long term non-progressor EC as defined by viral loads typically less than the LLD of commercially available assays and clinical and laboratory criteria (no OIs, no ART, stable CD4 T cell counts for more than 3 years). Viral load blips are allowed as long as they are less than 500 copies/mL and flanked by viral load measurements less than 100copies/mL. Viral load <100c/mL will be acceptable for eligibility at screening.
4. In women of childbearing potential, with no plans for pregnancy for the next 15 months and willing to use 2 investigator approved highly reliable methods of birth control consistently while on the study or in 3 month follow up.
5. Willingness to have samples stored for future research.
6. Not on a statin or ASA for the past 6 months.

ART <50 Arm

1. Age greater than or equal to 18 years.
2. Documented HIV-1 infection confirmed by enzyme-linked immunosorbent assay (ELISA) and Western blot tests.
3. In women of childbearing potential, with no plans for pregnancy for the next 15 months and willing to use 2 investigator approved highly reliable methods of birth control consistently while on the study or in 3 month follow up.
4. On continuous combination ART >4 years.
5. HIV RNA <50 copies/mL (or less than 40 or less than 48 copies/mL, depending on the lower limit of detection of the assay used; transient periods of low level (<300) detectable virus, blips, acceptable if isolated and followed by viral loads less than the lower limit of detection) >3 years and current HIV-RNA less than the LLD of the commercially available assay used. Subject will be rescreened if HIV is detectable at screening visit.
6. Willingness to have samples stored for future research.
7. Not on a statin or ASA for the past 6 months.

EXCLUSION CRITERIA

1. Diagnosis of cardiovascular disease or hypercholesterolemia (LDL cholesterol 190 mg/dL).
2. Known hypersensitivity or allergy to ATV or ASA, including a history of myositis or rhabdomyolysis with statin or ASA use.
3. Other contraindication for ASA or statin therapy (active liver disease, peptic ulcer disease, etc.).
4. Women who are lactating, pregnant, or actively trying to become pregnant or considering pregnancy over the likely span of the study (including women of childbearing potential who are unwilling to use adequate contraception throughout the study).
5. Any chronic inflammatory condition either requiring anti-inflammatory medication (systemic corticosteroids, daily NSAID use,immunomodulating medications) which may, in the opinion of the investigator, confound the interpretation of soluble inflammatory biomarkers. While on study, short term (less than 5 days) NSAID use will be allowed at the discretion of the investigator.
6. Active drug use or alcohol abuse that, in the opinion of the investigator, may interfere with the ability of the subject to participate in the study or that may unacceptably increase the risk of the study intervention..
7. Safety laboratory cut offs: coagulation (INR >2 upper limit of normal [ULN], PLT<75K), renal function (GFR<60), liver function (ALT or Alkaline phosphatase or direct bilirubin >2x ULN), aldolase <1.5 ULN and anemia (Hg <9 mg/dL).
8. Antiretroviral therapy with tipranivir, or any therapy which combines non-nucleoside reverse transcriptase inhibitors with protease inhibitors.
9. Chronic hepatitis C co-infection. However, if a subject has more than 24 weeks of sustained virologic response (SVR), the subject can be considered for eligibility.
10. If either MR or apheresis is contraindicated, subject may still participate without this procedure. In the case of missed apheresis, a 30 mL research blood draw will be substituted (see Appendices B and C).

    * If statin initiation is indicated per current guidelines, subject will be counseled to consult with their PMD. If the subject then chooses to take part in the study, we will provide their PMD with all pertinent lab results during the course of the study, if requested.

Co-enrollment Guidelines: Co-enrollment in other trials will be restricted, other than enrollment on observational studies. Study staff should be notified of co-enrollment as it may require the approval of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-04-18 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irini Sereti, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Hennipen County Medical Center, Minneapolis, Minnesota

REFERENCES:
- [Background] Deeks SG, Phillips AN. HIV infection, antiretroviral treatment, ageing, and non-AIDS related morbidity. BMJ. 2009 Jan 26;338:a3172. doi: 10.1136/bmj.a3172. No abstract available. PMID 19171560
- [Background] Krishnan S, Wilson EM, Sheikh V, Rupert A, Mendoza D, Yang J, Lempicki R, Migueles SA, Sereti I. Evidence for innate immune system activation in HIV type 1-infected elite controllers. J Infect Dis. 2014 Mar;209(6):931-9. doi: 10.1093/infdis/jit581. Epub 2013 Nov 1. PMID 24185941
- [Background] Funderburg NT, Mayne E, Sieg SF, Asaad R, Jiang W, Kalinowska M, Luciano AA, Stevens W, Rodriguez B, Brenchley JM, Douek DC, Lederman MM. Increased tissue factor expression on circulating monocytes in chronic HIV infection: relationship to in vivo coagulation and immune activation. Blood. 2010 Jan 14;115(2):161-7. doi: 10.1182/blood-2009-03-210179. Epub 2009 Oct 14. PMID 19828697
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-I-0039.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Daily Aspirin; Daily Lipitor: HIV Infected on ART
  HIV Infected off ART
Period: Overall Study
Arm/Group | Daily Aspirin | Daily Lipitor
Started | 26 | 27
Completed | 24 | 20
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Daily Aspirin; Daily Atorvastatin: HIV Infected on ART
  Elite controllers not on ART
- Total: Total of all reporting groups
Arm/Group | Daily Aspirin | Daily Atorvastatin | Total
Number analyzed (Participants) | 24 | 20 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [48.25 to 57.75] | 54 [40 to 58.75] | 54 [44 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 18 | 14 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 9 | 4 | 13
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 24 | 20 | 44
CD4 [Median (Inter-Quartile Range); unit: cells/μL] | 595 [485 to 826] | 717 [509 to 843] | 650 [500 to 840]
Total Cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 174 [160 to 203] | 173 [144 to 200] | 173 [150 to 202]
Hypertension [Count of Participants; unit: Participants] | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes in sCD14 After 9 Months of Treatment With Aspirin or Atorvastatin
Description: sCD14 change between baseline (average of month 0 and month 3 in the study) and month 12
Time Frame: Month 12
Measure: Median (95% Confidence Interval); unit: pg/mL
Arm/Group | Daily Aspirin | Daily Atorvastatin
Number analyzed (Participants) | 24 | 20
pg/mL | -0.131 [-0.417 to -0.032] | -0.09 [-0.528 to 0.22]
Statistical Analysis 1: Comparison: Daily Atorvastatin; Wilcoxon rank sum test was used to compare the change of sCD14 from baseline and month 12 measurement within each arm; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney) — Threshold for statistical significance was a priori set to <0.05
Statistical Analysis 2: Comparison: Daily Aspirin; Wilcoxon rank sum test was used to compare the change of sCD14 from baseline and month 12 measurement within each arm; Test type: Other; p = 0.022, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Changes in sCD14 in EC and ART <50 Groups Treated With Aspirin or Atorvastatin.
Description: sCD14 change between baseline (average of month 0 and month 3 in the study) and month 12
Time Frame: Month 12
Measure: Median (95% Confidence Interval); unit: pg/mL
Groups:
- Daily Aspirin on ART; Daily Atorvastatin on ART: Treated Individuals on Chronic Antiretroviral Therapy
- Daily Aspirin Not on ART; Daily Atorvastatin Not on ART: Elite controllers not on Chronic Antiretroviral Therapy
Arm/Group | Daily Aspirin on ART | Daily Aspirin Not on ART | Daily Atorvastatin on ART | Daily Atorvastatin Not on ART
Number analyzed (Participants) | 15 | 9 | 12 | 8
pg/mL | -0.1249 [-0.6963 to 0.1367] | -0.1353 [-0.417 to 0.005] | -0.3242 [-0.79 to -0.004] | 0.1758 [-0.17 to 0.698]
Statistical Analysis 1: Comparison: Daily Aspirin on ART; Wilcoxon rank sum test was used to compare the change of sCD14 from baseline and month 12 measurement within each arm; Test type: Other; p = 0.13, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Daily Aspirin Not on ART; Wilcoxon rank sum test was used to compare the change of sCD14 from baseline and month 12 measurement within each arm; Test type: Other; p = 0.097, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Daily Atorvastatin on ART; Wilcoxon rank sum test was used to compare the change of sCD14 from baseline and month 12 measurement within each arm; Test type: Other; p = 0.0269, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Daily Atorvastatin Not on ART; Test type: Other; p = 0.25, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Daily Aspirin on ART vs Daily Aspirin Not on ART vs Daily Atorvastatin on ART vs Daily Atorvastatin Not on ART; Test type: Other; Plasma biomarkers (CRP, sCD14, TF, IL-6) were log(e) transformed and a linear mixed effect model with the biomarker as outcome and with random slope per participant was used to calculate the percentage of change from baseline

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 3 months after the end of the drug.
Groups:
- Daily Aspirin; Daily Atorvastatin: HIV Infected on ART
  Elite controllers not on Chronic Antiretroviral Therapy
Arm/Group | Daily Aspirin | Daily Atorvastatin
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/24 | 1/23
Other Adverse Events (participants affected / at risk) | 12/24 | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Aspirin (N=24) | Daily Atorvastatin (N=23)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Aspirin (N=24) | Daily Atorvastatin (N=23)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gonorrhea (Infections and infestations) | 1 (1) | 0 (0)
White Blood Cell Decreased (Investigations) | 1 (1) | 0 (0)
Blood Creatinine Increase (Investigations) | 3 (3) | 0 (0)
Oesophageal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size, study was completed earlier compared to expected sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT02081638/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT02081638/ICF_001.pdf